CLINICAL TRIAL: NCT02626299
Title: Assessment of DHA On Reducing Early Preterm Birth (ADORE Trial)
Brief Title: Assessment of DHA On Reducing Early Preterm Birth
Acronym: ADORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Cincinnati (Other); Ohio State University (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Carlson, PhD, Professor, Dietetics and Nutrition, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00003455
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Early preterm birth; Very low birth weight; Low birth weight; Pregnancy outcome; Docosahexaenoic acid (DHA); Randomized cliinical trial; Superiority trial; Adaptive design
MeSH Terms: conditions — Premature Birth | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 200 mg/day DHA (Placebo Comparator): Participants will receive 2 placebo pills/day that do not contain DHA. Like the experimental group, they will be given a supplement of Docosahexaenoic acid - 200mg/day , a common amount in prenatal vitamins.
  Interventions: Drug: Docosahexaenoic acid - 200mg/day; Other: Placebo
- 1000 mg/day DHA (Experimental): The intervention includes Docosahexaenoic acid - 800mg/day per day provided in two 400 mg capsules. The intervention group as well as the active comparator group will be given 1-200 mg/capsule per day of DHA that is a common amount in prenatal vitamins.
  Interventions: Drug: Docosahexaenoic acid - 800mg/day; Drug: Docosahexaenoic acid - 200mg/day

INTERVENTIONS:
Drug: Docosahexaenoic acid - 800mg/day — All participants will take 1000 mg/DHA per day (1 capsule will be labeled with 200 mg; 2 capsules will be masked with 400 mg each)
  Other Names: DHA
  Arms: 1000 mg/day DHA
Drug: Docosahexaenoic acid - 200mg/day — The control group will receive 1-capsule containing 200 mg DHA/d.
  Other Names: DHA
Other: Placebo — Participants will receive 2 capsules (masked) containing half soybean oil and half corn oil equaling 800 mg.The soybean and corn oil combination does not contain DHA.
  Arms: 200 mg/day DHA

SUMMARY:
The purpose of this study is to determine if giving a larger amount of DHA than currently included in some prenatal supplements can reduce early preterm birth (birth before 34 weeks of pregnancy).

DETAILED DESCRIPTION:
Docosahexaenoic acid (DHA) is a nutrient found in some fish and eggs and its intake in US diets is typically low. Because DHA is important for early brain development, it has recently been added to many prenatal supplements. The usual amount is around 200 mg/day. Participants in this study are guaranteed to receive at least 200 mg/day of DHA.

Almost 5 in 100 births in the US occur before 34 weeks of pregnancy. There is no way to predict which births will occur before 34 weeks. In an earlier study conducted at the University of Kansas Medical Center, women who received 600 mg DHA/day compared to no DHA had fewer births before 34 weeks of pregnancy with fewer complications of preterm birth.

This study is designed to compare standard care (200 mg/day of DHA) to a higher amount of DHA (1000 mg/day) to determine if the higher amount will reduce early preterm birth (birth before 34 weeks of pregnancy). Individual participation in this study is expected last about 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females 18 years and older 12 to 20 weeks gestation at study entry
* Agree to consume study capsules and a typical prenatal supplement of 200 mg DHA
* Available by telephone
* Able to speak and read in either English or Spanish language

Exclusion Criteria:

* Expecting multiple infants
* Gestational age at baseline <12 weeks or >20 weeks
* Unable or unwilling to agree to consume capsules until delivery
* Unwilling to discontinue use of another prenatal supplement that contains greater than or equal to 200 mg DHA per day
* Women with allergy to any component of DHA product (including algae), soybean oil or corn oil

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of Early Preterm Birth (<34 weeks gestation) | Baseline to 34 Weeks
  Bayesian posterior mean and 95% credible interval of pregnancies which result in an early preterm birth (birth before 34 weeks of pregnancy) by DHA dose
Occurrence of Early Preterm Birth (<34 weeks gestation) | Baseline to 34 weeks
  Bayesian posterior mean and 95% credible interval of pregnancies which result in an early preterm birth (birth before 34 weeks of pregnancy) by DHA dose and DHA status at enrollment (low/high) (modified statistical analysis plan while study was underway)
Maternal and infant adverse and serious adverse events | Enrollment to 30 days past last birth
  Bayesian posterior mean and 95% credible interval by dose

SECONDARY OUTCOMES:
Very low birth weight | At birth
  Bayesian posterior mean and 95% credible interval <1500 grams by dose
Low birth weight | birth
  Bayesian posterior mean and 95% credible interval <2500 grams by dose
Maternal and infant DHA status | birth
  Bayesian posterior mean and 95% credible interval red blood cell phospholipid DHA (weight percent of total fatty acids) at enrollment and birth by dose
Gestational age | birth
  Bayesian posterior mean and 95% credible interval weeks gestation at birth by dose
Birth weight | birth
  Bayesian posterior mean and 95% credible interval in grams by dose
Length and head circumference | birth
  Bayesian posterior mean and 95% credible interval in centimeters by dose
Preterm birth (<37 weeks) | birth
  Bayesian posterior mean and 95% credible interval in weeks by dose
Preterm birth (<37 weeks) | birth
  Number of pregnancies ending in preterm birth by dose
Pre-eclampsia | 12-20 weeks gestation through birth at an average of 40 weeks
  Bayesian posterior mean and 95% credible interval
Pre-eclampsia | 12-20 weeks gestation through birth at an average of 40 weeks
  Number of patients with pre-eclampsia by dose
Gestational diabetes | 12-20 weeks gestation through birth at an average of 40 weeks
  Bayesian posterior mean and 95% credible interval by dose
Gestational diabetes | 12-20 weeks gestation through birth at an average of 40 weeks
  Number of patients with gestational diabetes by dose
Cesarean section | birth
  Bayesian posterior mean and 95% credible interval by dose
Cesarean section | birth
  Number of patients with c-section by dose
Spontaneous labor | birth
  Bayesian posterior mean and 95% credible interval by dose
Spontaneous labor | birth
  Number of patients with spontaneous labor by dose
Admissiion of neonate to a neonatal intensive care unit | birth
  Bayesian posterior mean and 95% credible interval by dose
Admissiion of neonate to a neonatal intensive care unit | birth
  Number of neonates admited to a neonatal intensive care unit by dose

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Carlson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Wang Y, Gajewski BJ, Valentine CJ, Crawford SA, Brown AR, Mudaranthakam DP, Camargo JT, Carlson SE. DHA, nutrient intake, and maternal characteristics as predictors of pregnancy outcomes in a randomised clinical trial of DHA supplementation. Clin Nutr. 2023 Nov;42(11):2229-2240. doi: 10.1016/j.clnu.2023.09.005. Epub 2023 Sep 20. PMID 37806075
- [Derived] Carlson SE, Gajewski BJ, Valentine CJ, Sands SA, Brown AR, Kerling EH, Crawford SA, Buhimschi CS, Weiner CP, Cackovic M, DeFranco EA, Mudaranthakam DP, Rogers LK. Early and late preterm birth rates in participants adherent to randomly assigned high dose docosahexaenoic acid (DHA) supplementation in pregnancy. Clin Nutr. 2023 Feb;42(2):235-243. doi: 10.1016/j.clnu.2023.01.009. Epub 2023 Jan 11. PMID 36680919
- [Derived] Mudaranthakam DP, Brown A, Kerling E, Carlson SE, Valentine CJ, Gajewski B. The Successful Synchronized Orchestration of an Investigator-Initiated Multicenter Trial Using a Clinical Trial Management System and Team Approach: Design and Utility Study. JMIR Form Res. 2021 Dec 22;5(12):e30368. doi: 10.2196/30368. PMID 34941552
- [Derived] Carlson SE, Gajewski BJ, Valentine CJ, Kerling EH, Weiner CP, Cackovic M, Buhimschi CS, Rogers LK, Sands SA, Brown AR, Mudaranthakam DP, Crawford SA, DeFranco EA. Higher dose docosahexaenoic acid supplementation during pregnancy and early preterm birth: A randomised, double-blind, adaptive-design superiority trial. EClinicalMedicine. 2021 May 17;36:100905. doi: 10.1016/j.eclinm.2021.100905. eCollection 2021 Jun. PMID 34308309
- [Derived] Carlson SE, Gajewski BJ, Valentine CJ, Rogers LK, Weiner CP, DeFranco EA, Buhimschi CS. Assessment of DHA on reducing early preterm birth: the ADORE randomized controlled trial protocol. BMC Pregnancy Childbirth. 2017 Feb 13;17(1):62. doi: 10.1186/s12884-017-1244-5. PMID 28193189